CLINICAL TRIAL: NCT01935635
Title: A Clinical Trial on Hepatitis B Vaccine Activated-DCs Combined With Peg-interferon or Nucleotide Analogs in Chronic Hepatitis B
Brief Title: A Clinical Trial on HB-Vac Activated-DCs Combined With Peg-IFN or NAs in CHB
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Ruijin Hospital (Other); Second People's Hospital of Yunnan Province (Other)
Responsible Party: Principal Investigator, Yuehua Huang, director of liver disease laboratory, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014ZX10002002-002
Record Dates: First submitted 2013-09-01; First posted 2013-09-05 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Chronic Hepatitis B
Keywords: CHB; Antiviral; Dentritic cells; Immune Therapy
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- HPDCs-T immune therapy combined with IFN (Experimental): HPDCs-T immune therapy:one time every 2 weeks during 12 weeks to 36 weeks, about 2*105-1*106 cells per time,total 12 times; IFN therapy (Peg-IFN α-2b/2a):one time every 1 week according to the standards for 48 weeks
  Interventions: Biological: HPDCs-T immune therapy
- HPDCs-T immune therapy combined with ETV (Experimental): HPDCs-T immune therapy:one time every 2 weeks during 12 weeks to 36 weeks, about 2*105-1*106 cells per time,total 12 times; Entecavir(ETV)therapy:0.5mg per day according guidelines for the treatment of chronic hepatitis B in the Asia Pacific Region
  Interventions: Biological: HPDCs-T immune therapy
- HPDCs-T immune therapy combined with LdT (Experimental): HPDCs-T immune therapy:one time every 2 weeks during 12 weeks to 36 weeks, about 2*105-1*106 cells per time,total 12 times; Telbivudine(LdT)therapy:600mg per day according guidelines for the treatment of chronic hepatitis B in the Asia Pacific Region
  Interventions: Biological: HPDCs-T immune therapy
- IFN treatment (No Intervention): IFN therapy (Peg-IFN α-2b/2a):one time every 1 week according to the standards for 48 weeks
- ETV treatment (No Intervention): Entecavir(ETV)therapy:0.5mg per day according guidelines for the treatment of chronic hepatitis B in the Asia Pacific Region
- LdT treatment (No Intervention): Telbivudine(LdT)therapy:600mg per day according guidelines for the treatment of chronic hepatitis B in the Asia Pacific Region

INTERVENTIONS:
Biological: HPDCs-T immune therapy — HPDCs-T immune therapy:one time every 2 weeks during 12 weeks to 36 weeks, IV (in the vein), about 2*105-1*106 cells per time,total 12 times;
  Other Names: The HBsAg sensitized dendritic cells activated T cells; HBsAg Pulse DCs-T
  Arms: HPDCs-T immune therapy combined with ETV; HPDCs-T immune therapy combined with IFN; HPDCs-T immune therapy combined with LdT

SUMMARY:
The purpose of this study is to investigate whether HB-Vac Activated-DCs Combined With Peg-IFN or NAs has more efficacy than Peg-IFN or NAs alone in the treatment of chronic hepatitis B patients

DETAILED DESCRIPTION:
The 450 patients meeting the entry criteria are divided into 6 groups, the clinical trial procedure is divided into 3 parts, according to the following steps:

Part1 (0-12W):

1. The research objects will be grouped according to the principle of a multicenter, randomized, open, parallel controlled clinical trial, 300 cases of cell therapy groups (100 cases with PEG-IFN treatment, LdT treatment for 100 cases, ETV treatment for 100 cases), 150 cases of control groups (PEG-IFN therapy in 50 cases, LdT therapy for 50 cases, ETV treatment for 50 cases).

   Part2 (12-36W):
2. Cell therapy groups: enter the HBsAg sensitized dendritic cells activated T cells (HBsAg Pulse DCs-T, HPDCs-T) immune therapy combined with interferon (IFN) or nucleoside analogues treatment (NAs), infusion of HPDC-T every 2 weeks for 1 time, total 12 times.
3. Control groups: antiviral therapy used only (IFN or NAs).

   Part3 (36-72W):
4. The observation stage: discontinuation of interferon in the treatment of 48 weeks; NAs cases will continue on treatment with NAs.

HPDCs-T produced procedure:

The first step: 1-7 days Monocytes will be isolated from peripheral blood of patients. The monocytes obtained will be then incubated in fresh serum-free AIM-V medium (Gibco) containing 800U/ml of GM-CSF and 400U/ml of IL-4 (Peprotech) for 5 days. After 5 days of culture in vitro, The DCs induced will be cultured with a commercially available hepatitis B vaccine containing 10 ug of HBsAg (GSK) for 2 days.

The second step: 8-14 days The hepatitis B vaccine sensitized DCs (HPDCs) (from the first step) will be sub-cultured with patient's own PBMCs for 7 days: HBsAg can be efficiently presented to PBMCs by DCs, with producing HBV specific CTLs and HTLs (HPDCs-T).

The third step: 15 days The PBMCs (the second step) containing enough HPDCs-T will be transfused back into the patient.

ELIGIBILITY:
Inclusion Criteria:

serum hepatitis B surface antigen(HBsAg) positive for at least 6 months; HBV DNA loads≥ 104IU/ml(Roche Cobas); Containing the IFN treatment: 2ULN ≤ ALT ≤ 10ULN and TBil ≤ 2ULN; Containing the ETV/LdT treatment: 2ULN ≤ ALT and TBil ≤ 5ULN; All patients have not received antiviral treatment or immunotherapy for the last 6 months.

Exclusion Criteria:

superinfection or co-infection with hepatitis A, C, D, E, cytomegalovirus and HIV, or Epstein-Barr virus; other liver diseases such as alcoholic liver disease, drug-induced hepatitis, Wilson disease and autoimmune hepatitis; ascites or gastrointestinal bleeding or peptic ulcer or esophageal varix by electronic gastroscope examination; liver cirrhosis; severe bacterial or fungal infections; a history of diabetes or cardiac disease or hypertension or nephrosis; pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2015-01; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
HBV makers | 01/01/2014-31/12/2016, total 6 times (3 years)
  HBV DNA loads,HBsAg/HBsAb titer,HBeAg/HBeAb titer

SECONDARY OUTCOMES:
Coagulation tests | 01/01/2014-31/12/2016, total 6 times (3 years)
  PT,PTA,INR
liver function | 01/01/2014-31/12/2016, total 6 times (3 years)
  ALT,AST,Tbil,Alb
alpha-fetal protein | 01/01/2014-31/12/2016, total 4 times (3 years)
  AFP;Biomarkers of hepatocellular carcinoma,one time every 24 weeks
B ultrasound or MRI examination of the liver | 01/01/2014-31/12/2016, total 2 times (3 years)
  The examination is performed both at the end of the pre-experiment and the main experiment
Liver biopsy | 01/01/2014-31/12/2016, total 2 times (3 years)
  The examination is performed both before and during experiment.

CONTACTS AND LOCATIONS:
Overall Officials: Yuehua Huang, Doctor, Study Director — Deparment of Infectious Diseases, the Third Affiliated Hospital of Sun Yat-sen University
Locations (3):
- China (3):
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The second people's hospital of yunnan province, Kunming, Yunnan
  - Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gu Y, Gu L, Chen L, Li J, Liao C, Bi Y, Huang Z, Cai W, Wei J, Huang Y. Immunotherapy Using HBV Vaccine Pulsed DCs and Induced T-Cells Combined Antiviral Drugs in Treatment Naive CHB Patients-A Multi-Centre Phase II Study. J Viral Hepat. 2025 Feb;32(2):e14045. doi: 10.1111/jvh.14045. PMID 39815989